CLINICAL TRIAL: NCT00561977
Title: Finding a Simple Message to Improve Dietary Quality for Cancer and Heart Disease
Brief Title: Cancer Dietary Objectives Study
Acronym: CanDo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Barbara Olendzki, Nutrition Program Director, UMass Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRG 93-033
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Results first posted 2011-09-02 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Cancer; Heart Disease
Keywords: Nutrition; Dietary Quality; Weight loss
MeSH Terms: conditions — Neoplasms; Heart Diseases; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Fiber Diet (Active Comparator): high fiber diet (≥30 grams of total fiber per day); reduction of calories to -500 from resting metabolic rate (RMR), not less than 1200 kcal per day.
  Interventions: Behavioral: High Fiber Diet
- Low Saturated Fat (Active Comparator): low saturated fat diet (≤7% of total calories); -500 calories from RMR, not less than 1200 kcal per day.
  Interventions: Behavioral: low saturated fat diet
- Combination Diet (Active Comparator): Combination low saturated fat (≤7% of total calories);high fiber (>30g fiber per day) -500 kcal from RMR, not less than 1200 kcal/day.
  Interventions: Behavioral: Combination diet

INTERVENTIONS:
Behavioral: High Fiber Diet — high fiber diet (≥30 grams of total fiber per day); reduction of calories to -500 from resting metabolic rate (RMR), not less than 1200 kcal per day.
  Arms: High Fiber Diet
Behavioral: low saturated fat diet — low saturated fat diet (≤7% of total calories); -500 calories from RMR, not less than 1200 kcal/day.
  Arms: Low Saturated Fat
Behavioral: Combination diet — combination low saturated fat high fiber diet, with calorie restriction as specified.
  Arms: Combination Diet

SUMMARY:
We hypothesize that adding beneficial high fiber foods to the diet will result in better overall dietary quality (measured by the Alternate Healthy Eating Index), which has been shown to be associated with cancer, than either reducing saturated fat, or a combination of high fiber and low saturated fat.

DETAILED DESCRIPTION:
Summary of Grant:

Several studies have demonstrated that poor dietary quality is associated with obesity and certain cancers, such as gastrointestinal, colorectal, and hormonal cancers. Dietary interventions aimed at improving diet are plagued by poor adherence, possibly due to the complexity of changing multiple diet components. Complex public health messages are associated with worse adherence and reduced capacity to impact health outcomes. If a simple public health recommendation for diet was effective at changing multiple aspects of diet, adherence and impact could be maximized. However, research has yet to test which single dietary message has the greatest impact on overall diet quality, and consequently, potential for cancer and heart disease prevention. Thus far, dietary interventions have tested varying combinations of multiple recommendations; however, a single dietary recommendation may have a synergistic beneficial effect on other areas of diet, precluding the need to make the message overly complex.

The present study compares 3 dietary change conditions that are hypothesized to have high potential for synergistic effects on other unaddressed areas of diet, and consequently overall dietary quality. Patients were randomized to one of three arms:

1. low saturated fat diet (≤7% of total calories);
2. high fiber diet (≥30 grams of total fiber per day);
3. combination arm: low saturated fat and high fiber.

Each participant was instructed to reduce calories by -500 kcal/day from his/her resting metabolic rate (RMR), but total calories was not less than 1200 calories per day.

Additionally, Dr. Ira Ockene, professor of medicine, director of preventive cardiology program, generously offered to pay for blood draws and blood lipids and glucose analysis at each visit to make the study valuable from both cancer and heart disease research perspectives.

Specific aims:

1. Develop intervention materials. Intervention materials that specifically aid participants towards a low saturated fat or high fiber diet, or combination change developed for each condition.
2. Preliminary test of intervention. We will calculate change in diet quality, lipids, body weight, waist circumference, and blood pressure at 3- and 6-months. We hypothesize that the single change conditions will produce more changes than the complex condition and that adding beneficial high fiber foods to the diet will result in improved dietary quality (measured by the Alternative Healthy Eating Index) than reducing saturated fat. Secondary outcomes include calorie intake, micro- and macronutrients at baseline, physical activity, and observe changes at 3- and 6-months.
3. Adherence. We will examine adherence to the treatment protocol so that appropriate adjustments to the intervention can be made, if necessary, to enhance adherence in the larger randomized clinical trial.
4. Data for sample size estimation. We will document means and standard deviations on measures so that sample size can be estimated for the larger randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. BMI ≥25, and ≤40.
2. >=21 years of age, less than 81 years of age.
3. has primary care physician's approval to participate in all aspects of the study,
4. speaks, reads, and understands English at 6th grade level minimum
5. residing in local area for the duration of the study.
6. available for bi-monthly sessions (6 individual nutrition counseling visits)

Exclusion Criteria:

1. presence of a psychological disorder that will limit his/her ability to participate (such as an eating disorder, uncontrolled bipolar disorder)
2. unwilling to provide informed consent
3. presence of unstable medical disorder (e.g., uncontrolled hypertension, uncontrolled diabetes, etc), or a medical disorder associated with a life expectancy less than 2 years.
4. currently taking any medication known to affect weight or appetite
5. smokes more than 3 cigarettes a day on average
6. Has a dietary restriction that precludes changing to the healthy diet, i.e.; Crohn's disease, ulcerative colitis, renal disease, active diverticulitis, etc.
7. currently following a specific diet plan (low saturated fat/meat, or high fiber)
8. does not have a telephone
9. Pregnant, or planning to become pregnant (participant will be asked this question in telephone screening. If the participant becomes pregnant, they are asked to inform the principal investigator)
10. Has an active drug or alcohol problem within the past year -

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-05; Primary Completion 2008-05 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara C Olendzki, RD MPH, Principal Investigator — UMass Medical School
Locations (1):
- UMass Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Result] Olendzki BC, Ma Y, Schneider KL, Merriam P, Culver AL, Ockene IS, Pagoto S. A simple dietary message to improve dietary quality: Results from a pilot investigation. Nutrition. 2009 Jul-Aug;25(7-8):736-44. doi: 10.1016/j.nut.2009.01.009. Epub 2009 Apr 9. PMID 19359142

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 78 patients responding to advertisements at UMass Medical School intranet, 36 (41%) eligible overweight and obese patients were consented to participate in the study. Dates of recruitment were May-August 2007.
Pre-assignment Details: 23 ineligible, 5 refused screening, 12 patients put on waiting list, 2 patients dropped prior to randomization due to pregnancy. 2 patients added from waiting list to active participation.
Period: Overall Study
Arm/Group | High Fiber Diet | Low Saturated Fat | Combination Diet
Started | 12 | 12 | 12
Completed | 12 | 9 | 10
Not Completed | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Pregnancy | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Fiber Diet | Low Saturated Fat | Combination Diet | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 12 | 35
  >=65 years | 0 | 1 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 48.42 (9.77) | 53.00 (12.5) | 41.33 (15.89) | 47.58 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 10 | 31
  Male | 1 | 2 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Dietary Quality
Description: Dietary quality was measured by the Alternative Healthy Eating Index (AHEI), a scale of healthy eating that goes from zero to 80 (best score).
Time Frame: 6 mos
Measure: Mean (Standard Deviation); unit: score
Arm/Group | High Fiber Diet | Low Saturated Fat | Combination Diet
Number analyzed (Participants) | 12 | 9 | 10
score | 38.78 (3.20) | 41.18 (3.51) | 39.76 (3.70)
Statistical Analysis 1: Comparison: High Fiber Diet vs Low Saturated Fat vs Combination Diet; Mean dietary quality score by visit and study group was estimated using SAS PROC MIXED. All analyses were performed using SAS 9.13 (SAS Institute, Cary, NC, USA); Test type: Superiority or Other; p = 0.14, Mixed Models Analysis; time measurement, treatment group, interaction between time and group term as fixed effect, subject as random effect

2. Primary Outcome: Dietary Quality, Possible Score From Zero to 80 (Best Quality Diet).
Description: The AHEI consists of 8 components (eg, vegetables,trans fat). Each contributed 0-10 points to the total score; a score of 10 indicates that the recommendations were fully met, whereas a score of 0 represents the least healthy dietary behavior. Intermediate intakes were scored proportionately between 0 and 10. All component scores were summed to obtain a total AHEI score ranging from zero(worst) to 80(best).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score
Arm/Group | High Fiber Diet | Low Saturated Fat | Combination Diet
Number analyzed (Participants) | 12 | 9 | 10
score | 44.90 (3.51) | 44.90 (3.20) | 43.75 (3.70)

3. Secondary Outcome: Change in Weight From Baseline to 3 Months
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | High Fiber Diet | Low Saturated Fat | Combination Diet
Number analyzed (Participants) | 12 | 9 | 10
pounds | -7.0 (2.0) | -9.1 (2.2) | -6.7 (2.3)

4. Secondary Outcome: Change in Weight From Baseline to 6 Months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | High Fiber Diet | Low Saturated Fat | Combination Diet
Number analyzed (Participants) | 12 | 9 | 10
pounds | -9.1 (2.0) | -10.2 (2.2) | -7.0 (2.3)

5. Secondary Outcome: Change in Calories From Baseline to 3 Months
Description: kilocalories
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: calories
Arm/Group | High Fiber Diet | Low Saturated Fat | Combination Diet
Number analyzed (Participants) | 12 | 9 | 10
calories | -464.05 (94.52) | -190.90 (103.54) | -638.91 (109.15)

6. Secondary Outcome: Change in Calories From Baseline to 6 Months
Description: kilocalories
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: calories
Arm/Group | High Fiber Diet | Low Saturated Fat | Combination Diet
Number analyzed (Participants) | 12 | 9 | 10
calories | -364.82 (94.52) | -187.19 (103.54) | -626.32 (109.15)

ADVERSE EVENTS:
Arm/Group | High Fiber Diet | Low Saturated Fat | Combination Diet
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 1/12 | 0/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Fiber Diet (N=12) | Low Saturated Fat (N=12) | Combination Diet (N=12)
loss of consciousness from blood draw (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No